CLINICAL TRIAL: NCT03654690
Title: eTest: Real-time, Remote Monitoring System for Home-based HIV Testing Among High-risk Men Who Have Sex With Men
Acronym: eTest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Southern California (Other); The Miriam Hospital (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1804002021; 1R01MH114891-01A1 (NIH)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are not informed of their condition assignment, but may infer it via the procedures they are provided. Both investigators and staff assessing outcomes are blinded to participants' group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control (No Intervention): Participants will receive SMS text message reminders to get tested for HIV in a clinic.
- Standard Self-Testing (Active Comparator): Participants will receive an HIV self-test kit in the mail with no standardized follow-up from counselors.
  Interventions: Diagnostic Test: HIV self-test
- Enhanced Self-Testing (Experimental): Participants will receive an HIV self-test kit and will be contacted via telephone for counseling within 24 hours of opening their test.
  Interventions: Diagnostic Test: HIV self-test; Behavioral: Counseling

INTERVENTIONS:
Diagnostic Test: HIV self-test — Home delivery of HIV self-test kits (OraSure OraQuick Rapid HIV test)
  Arms: Enhanced Self-Testing; Standard Self-Testing
Behavioral: Counseling — Post-Test HIV Risk ReductionCounseling
  Arms: Enhanced Self-Testing

SUMMARY:
The proposed research will conduct a fully-powered efficacy trial of this approach in areas with large populations of AA and H/L MSM and high HIV incidence: Jackson, MS, Los Angeles, CA, and Boston, MA. High-risk MSM who have not tested for HIV in the last year will be recruited from MSM-oriented "hook-up" mobile apps, and assigned to receive either (1) HBST with post-test phone counseling/referral ("eTEST" condition), (2) "standard" HBST without active follow-up, or (3) reminders to get tested for HIV at a local clinic ("control" condition) at three month intervals over the course of 12 months. The investigators will explore the impact of the eTEST system on key outcomes, including rates of HIV testing, receipt of additional HIV prevention services, and PrEP initiation, compared with standard HBST or clinic-based testing reminders alone. The investigators will also explore the cost effectiveness of the eTEST system under various scenarios compared with relying on traditional, clinic-based testing alone.

DETAILED DESCRIPTION:
HIV disproportionately affects men who have sex with men (MSM) in the United States, and new infections continue to increase particularly among African American (AA) and Hispanic/Latino (H/L) MSM. Past studies estimate that up to 50% of these new infections originate from the approximately 20% of MSM who are unaware of their status. Expanded HIV testing can produce reductions in incidence when implemented on a broad scale by facilitating earlier diagnosis and treatment. Rates of HIV testing are particularly low among AA and H/L MSM, and innovative approaches to encourage testing may help address high incidence in these men. Home-based, self-testing (HBST) for HIV offers considerable promise for increasing the number of MSM who are aware of their status by overcoming key barriers to clinic-based testing, such as inconvenience and confidentiality concerns. HBST may also be particularly well-suited for AA and H/L MSM, given that stigma and mistrust of medical care contribute to low testing rates. Despite its promise, however, many are concerned that HBST does not sufficiently connect users with critical post-testing resources, such as confirmatory testing and care among those who test positive, and that these limitations may result in delayed linkage to care. Existing, FDA-approved HBST kits provide a free, 24-hour helpline that offers these services to those who seek it, but few users do, and this "passive" approach may miss critical opportunities to engage with MSM for further prevention services.

To address these challenges, the investigators developed a mobile health platform ("eTEST") that uses internet-of-things (IoT) technologies to monitor when HBST users open their tests in real time, allowing the investigators to provide timely, "active" follow-up counseling and referral over the phone after they do so. In a pilot study, the investigators show that providing HBST by mail at regular intervals boosted rates of any/repeat HIV testing among high-risk MSM compared with clinic-based testing reminders. Moreover, those who received follow-up phone counseling after HBST were more likely to receive risk reduction counseling, to consult with a medical provider about PrEP, and to initiate PrEP. Given these promising results, the proposed research will conduct a fully-powered efficacy trial of this approach in areas with large populations of AA and H/L MSM and high HIV incidence: Jackson, MS, Los Angeles, CA, and Boston, MA. High-risk MSM who have not tested for HIV in the last year will be recruited from MSM-oriented "hook-up" mobile apps, and assigned to receive either (1) HBST with post-test phone counseling/referral ("eTEST" condition), (2) "standard" HBST without active follow-up, or (3) reminders to get tested for HIV at a local clinic ("control" condition) at three month intervals over the course of 12 months. The investigators will explore the impact of the eTEST system on key outcomes, including rates of HIV testing, receipt of additional HIV prevention services, and PrEP initiation, compared with standard HBST or clinic-based testing reminders alone. The investigators will also explore the cost effectiveness of the eTEST system under various scenarios compared with relying on traditional, clinic-based testing alone.

ELIGIBILITY:
Inclusion Criteria:

* report any of the following in the past six months: anal sex without condoms outside of a monogamous partnership with a recently tested, HIV-negative male, having been diagnosed with an STI, or being in an ongoing sexual partnership with an HIV-positive male
* not tested for HIV in the last 12 months
* have a stable residence in one of the site metros where they can securely receive packages
* use an iOS/Android smartphone with a data plan or home wifi
* fluent in either English or Spanish

Exclusion Criteria:

* currently on PrEP

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler B Wray, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the final dataset for this research has been assembled, the Project Coordinator will create an archival copy (which will contain no personally identifying information) to store, along with an electronic version of the codebooks of the study. Versions will be available in English, and outside investigators will be able to utilize the data by contacting the PIs and describing their purpose for using the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the publication of primary analyses. Data will be available for as long as requests are made.
Access Criteria: De-identified individual participant data will be available to outside investigators after the primary analyses have been conducted and are published.

REFERENCES:
- [Derived] Wray TB, Chan PA, Klausner JD, Mena LA, Brock JB, Simpanen EM, Ward LM, Chrysovalantis S. eTest: a limited-interaction, longitudinal randomized controlled trial of a mobile health platform that enables real-time phone counseling after HIV self-testing among high-risk men who have sex with men. Trials. 2020 Jul 16;21(1):654. doi: 10.1186/s13063-020-04554-1. PMID 32677999

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Started | 271 | 265 | 275
Completed | 270 | 265 | 275
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing | Total
Number analyzed (Participants) | 270 | 265 | 275 | 810
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.4) | 34.6 (12.6) | 35.2 (12.3) | 34.7 (12.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 269 | 258 | 268 | 795
  Trans/Other gender identity | 1 | 7 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 84 | 98 | 277
  Not Hispanic or Latino | 175 | 181 | 177 | 533
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 3 | 7
  Asian | 25 | 24 | 23 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 21 | 33 | 31 | 85
  White | 179 | 169 | 172 | 520
  More than one race | 20 | 16 | 23 | 59
  Unknown or Not Reported | 23 | 20 | 22 | 65
Region of Enrollment [Number; unit: participants]
  United States | 270 | 265 | 275 | 810

OUTCOME MEASURES:

1. Primary Outcome: Model Adjusted Probability of Any HIV Testing
Description: We used logistic regression with dummy-coded condition assignment as a predictor to test differences in outcomes across experimental conditions. A dummy-coded covariate indicating whether participants reported testing fewer than three times in the 3 years prior to enrolling was included in all models of HIV testing.
  We fit longitudinal mixed effects models for two outcomes, HIV testing and high-risk CAS events within a given follow-up period, given that these outcomes varied within participants across the study period. We specified distributions appropriate for each outcome (logistic for HIV testing and negative binomial for high-risk CAS events) with suitable link functions, unstructured covariance structures and robust standard errors. Time was included as a continuous covariate. A covariate reflecting pre-enrolment HIV testing and baseline CAS events were included in these models. We used an intent-to-treat approach for all analyses. Missing data were considered missing at random.
Time Frame: 12 month study period
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Number analyzed (Participants) | 270 | 265 | 275
percent probability | 57.0 [51.0 to 62.9] | 91.0 [87.9 to 94.6] | 89.4 [86.2 to 93.3]

2. Primary Outcome: Model Adjusted Probabilities of Repeat HIV Testing (>1)
Description: as for outcome 1
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Number analyzed (Participants) | 270 | 265 | 275
percent probability | 31.3 [25.7 to 36.9] | 79.4 [74.5 to 84.3] | 80.4 [75.7 to 85.1]

3. Primary Outcome: HIV Diagnoses
Description: count of participants who were ultimately diagnosed with HIV during the course of the study
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Number analyzed (Participants) | 270 | 265 | 275
Participants | 0 | 4 | 4

4. Secondary Outcome: Model Predicted Probability of Receipt of a Prescription for Pre-exposure Prophylaxis (PrEP)
Description: We used logistic regression with dummy-coded condition assignment as a predictor to test differences in outcomes across experimental conditions. A binary variable reflecting whether participants had ever had a PrEP prescription in the past was included for the PrEP prescription model. We specified two-way interactions between these covariates and condition assignment in all models, but none were significant and were excluded.
Time Frame: 12 month study period
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Number analyzed (Participants) | 270 | 265 | 275
percent probability | 20 [15 to 25] | 15 [10 to 19] | 15 [10 to 19]

5. Secondary Outcome: Model Predicted Probability of Receipt of Testing for Other Sexually-transmitted Infections
Description: We used logistic regression with dummy-coded condition assignment as a predictor to test differences in outcomes across experimental conditions. A dummy-coded covariate indicating whether participants reported testing fewer than three times in the 3 years prior to enrolling was included in all models of HIV testing. A similar covariate for STI testing was included in the STI testing model. We specified two-way interactions between these covariates and condition assignment in all models, but none were significant and were excluded.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Number analyzed (Participants) | 270 | 265 | 275
percent probability | 46 [40 to 52] | 49 [43 to 55] | 50 [44 to 56]

6. Other Pre Specified Outcome: Average Predicted Number of High-risk Casual Anal Sex (CAS) Events With Partners of Unknown HIV and PrEP Status
Description: We used logistic regression with dummy-coded condition assignment as a predictor to test differences in outcomes across experimental conditions. We specified two-way interactions between these covariates and condition assignment in all models, but none were significant and were excluded. We fit longitudinal mixed effects models for two outcomes, HIV testing and high-risk CAS events within a given follow-up period, given that these outcomes varied within participants across the study period. We specified distributions appropriate for each outcome (logistic for HIV testing and negative binomial for high-risk CAS events) with suitable link functions, unstructured covariance structures and robust standard errors. Time was included as a continuous covariate. A covariate reflecting pre-enrolment HIV testing and baseline CAS events were included in these models.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
Number analyzed (Participants) | 270 | 265 | 275
events | 2.03 [0.5 to 3.6] | 2.01 [0.5 to 3.5] | 1.46 [.3 to 2.6]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Control | Standard Self-Testing | Enhanced Self-Testing
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/265 | 0/275
Serious Adverse Events (participants affected / at risk) | 0/270 | 0/265 | 0/275
Other Adverse Events (participants affected / at risk) | 0/270 | 0/265 | 0/275

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03654690/Prot_SAP_002.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03654690/ICF_003.pdf